CLINICAL TRIAL: NCT06707532
Title: The Use of Muscle Relaxants During Electroporation Ablation (PFA) as a Potential Protective Factor Against Damage to Transverse Striated Muscle Tissue and the Heart
Brief Title: The Potential Protective Effect of Using Muscle Relaxants During Electroporation Ablation (PFA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 4th Military Clinical Hospital with Polyclinic, Poland (Other)
Responsible Party: Principal Investigator, Marek Szamborski, Medical Doctor, 4th Military Clinical Hospital with Polyclinic, Poland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 4_2024
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Kidney Failure, Acute; Myopathy; Drugs; Heart Arrhythmia; Succinylcholine Sensitivity; Muscle Relaxation; General Anesthetic Drug Adverse Reaction; Projection
Keywords: electroporation ablation (PFA); muscle relaxants; rocuronium; chronic pain; acute kidney failure; chronic heart failure; drug protection
MeSH Terms: conditions — Acute Kidney Injury; Myotoxicity; Arrhythmias, Cardiac; Butyrylcholinesterase deficiency; Muscle Hypotonia; Chronic Pain | interventions — Propofol; Anesthesia, General; Rocuronium

STUDY DESIGN:
Intervention Model Description: The subjects will be randomly divided into 2 groups. Group I will consist of patients undergoing general anaesthesia without the use of the muscle relaxant rocuronium during electric current application. Group II will consist of patients undergoing general anaesthesia with the muscle relaxant rocuronium. A total of 32 patients were initially planned for the study (16 patients in each of the two groups).
Who Masked: Participant, Care Provider
Masking Description: Before the procedure, the anaesthetist will be given a sealed envelope by a person unrelated to the project (hospital administrative staff), with a randomised method of anaesthesia based on simple randomisation. Before the procedure, each patient will have a transthoracic cardiac ultrasound (TTE). The patient will not know which study group he/she has been classified into. The operator performing the procedure will not be informed about the type of anaesthesia performed -[randomisation by double-blinding].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (no muscular relaxant) (Active Comparator): Group I - 16 patients undergoing general anaesthesia with endotracheal intubation, during the induction of anaesthesia, the patients will be administered a muscle relaxant from the depolarising group (Chlorsuccilin®) for the endotracheal intubation procedure (using precurarisation). This is a method of pharmacologically preventing the muscle fasciculations characteristic of depolarising agents. For this purpose, a low-dose muscle relaxant from the non-depolarising group - (rocuronium, Esmeron®) will be administered just before the actual dose of the depolarising agent. No muscle relaxant will be used during the actual procedure, but the level of muscle relaxation will be continuously monitored through the use of the NMT - TOF % technique (a method of measuring neuromuscular excitability that allows real-time assessment of muscle strength).
  Interventions: Drug: Propofol
- Group II (muscular relaxant) (Active Comparator): Group II -16 patients undergoing general anaesthesia with endotracheal intubation, during the induction of anaesthesia the patients will be administered a muscle relaxant from the depolarising group (rocuronium, Esmeron®) for the endotracheal intubation procedure (using precurarisation). This is a method of pharmacological prevention of muscle fasciculation, characteristic of depolarising agents. For this purpose, a low-dose muscle relaxant from the non-depolarising group (rocuronium, Esmeron®) will be administered just before the actual dose of the depolarising agent. During the procedure itself, the level of relaxation will be continuously monitored by using the NMT - TOF % technique (a method of measuring neuromuscular excitability that allows real-time assessment of muscle strength). During the ablation performed, the patient will be under the influence of a muscle relaxant from the non-depolarising group (rocuronium, Esmeron®).
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Propofol — Induction of anaesthesia:
  * Fentanyl 1-3ug/kg/m.c i.v.
  * Ketamine 50mg i.v.
  * Propofol 1.5-2mg/kg/m.c i.v.
  * Rocuronium 5mg (b.w.<60kg) 10mg (b.w.>60kg) i.v. Precurarisation
  * Chlorucinylcholine 1-1.5mg/kg/m.c i.v. -> Intubation
  Application (cycle of 5 pulses with 2000V biphasic alternating current) - during PFA:
  - In case of ventilatory distress pPeak >30 cm H2O ad hoc Propofol 0.25-0.75mg/kg/m.c i.v.
  Elimination of neuromuscular blockade:
  - To exclude residual relaxation after pre-curative: 1mg Atropine i.v. + 0.5mg Neostigmine i.v.
  Other Names: no muscular relaxant; general anaesthesia
  Arms: Group I (no muscular relaxant)
Drug: Rocuronium — Induction of anaesthesia:
  * Fentanyl 1-3ug/kg/m.c i.v.
  * Ketamine 50mg i.v.
  * Propofol 1.5-2mg/kg/m.c i.v.
  * Rocuronium 5mg (b.w.<60kg) 10mg (b.w.>60kg) i.v. Precurarisation
  * Chlorucinylcholine 1-1.5mg/kg/m.c i.v. -> Intubation
  Application (cycle of 5 pulses with 2000V biphasic alternating current) - during PFA:
  - rocuronium 0.1-0.3mg/kg/m.c i.v. For TOF <2
  Abolition of neuromuscular blockade:
  - Atropine 1-1.5mg i.v. + 1-3mg Neostigmine i.v. Or Sugammadex 2-4mg/kg/m.c i.v.
  Other Names: muscular relaxant; general anaesthesia
  Arms: Group II (muscular relaxant)

SUMMARY:
The study aims to improve the safety of the electroporation ablation (PFA) procedure by using muscle relaxants to reduce skeletal muscle damage during the procedure. It will also assess myocardial damage to improve the procedure's quality and speed up recovery after the procedure.

DETAILED DESCRIPTION:
The procedure of electroporation (PFA) is a method of atrial fibrillation ablation introduced in Poland in 2022. A biphasic high voltage current (2000 volts) is applied to the electrode placement site. Local coagulation of the site is followed by myocardial scarring and interruption of the pathological conduction pathway of premature electrical impulses in the heart. The patient, once qualified by the cardiologist for the procedure of electroporation ablation (PFA), will undergo a standard anaesthetic qualification process with assessment of basic demographics, comorbid conditions, medications taken, determination on the surgical risk scale.

Participants will be randomized into 2 groups. Group I will consist of patients undergoing general anaesthesia without the muscle relaxant rocuronium. Group II will consist of patients undergoing general anaesthesia with the muscle relaxant rocuronium. A total of 32 patients were initially planned for the study (16 patients in each of the two groups). Before the procedure, the anaesthetist will be given a sealed envelope by a person unrelated to the project (hospital administration staff) with a randomised method of anaesthesia based on simple randomisation. Before the procedure, each patient will have a transthoracic ultrasound of the heart (TTE). The patient will not know which study group he/she has been assigned to. The operator performing the procedure will not be informed about the type of anaesthesia used [double blind randomisation].

ELIGIBILITY:
Inclusion Criteria:

* Patients with requirement for PFA ablation for cardiac indications and ability to provide informed consent for study participation

Exclusion Criteria:

* Patients with allergies to the general anaesthetics used, genetic diseases of the neuromuscular plateau - e.g. Duchenne dystrophy, myasthenia gravis - and patients who do not gived informed consent to participate in the study will be excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Baseline laboratory parameters and additional tests | up to 24 hours before procedure
  Serum creatinine Serum potassium General morphology evaluation of HGB and PLT values Assessment of QoR-15 Measurement of heart size and mass on TTE ultrasound
During the procedure (before the start of current application) | before the start of current application
  Serum myoglobin Serum troponin Serum CPK
Endline laboratory parameters and additional tests | 12 hours after procedure
  Serum myoglobin Serum troponin Serum CPK Serum creatinine Serum potassium Total morphology evaluation of HGB and PLT values
NRS | Checked before procedure and every 6 hours for the first 24 hours after the procedure
  numerical pain scale 0-10 points
QoR - 15 | Administered to the patient before surgery and 24 hours after surgery
  post-operative quality of life and improvement scale 0-150 points

SECONDARY OUTCOMES:
BMI | Before performing procedure
  Body mass index 15-45

CONTACTS AND LOCATIONS:
Overall Officials: Marek Szamborski, MD, Principal Investigator — Senior Assistant
Locations (1):
- 4th Military Clinical Hospital with Polyclinic, Wroclaw, Lower Silesian Voivodeship, Poland